CLINICAL TRIAL: NCT04001478
Title: Non-invasive Testing for the Diagnosis of Early Oesophageal Cancer and Barrett's Dysplasia
Brief Title: Non-invasive Testing for Early oEesophageal Cancer and Dysplasia
Acronym: NEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Guts UK (Other); University College London Hospitals (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Northern Care Alliance NHS Foundation Trust (Other); London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19/LO/0780
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Oesophageal Cancer; Barrett Esophagus; Barretts Esophagus With Dysplasia
Keywords: Oesophageal Cancer; Barretts Esophagus with Dysplasia
MeSH Terms: conditions — Esophageal Neoplasms; Barrett Esophagus | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Patients who are attending hospital for a gastroscopy as part of their routine clinical care as a 2 week wait rule referral and those on Barrett's surveillance , will be asked to give a sample of their breath prior to the procedure.
  Interventions: Diagnostic Test: Breath test
- Early oesophageal cancer (T1)/ Barrett's high grade dysplasia: Patients who have known pre-diagnosed T1 oesophageal adenocarcinoma or HGD attending hospital as part of their clinical care will be asked to give a breath sample prior to their endoscopy resection/ cancer operation. Patients will be sampled upon return for follow up endoscopy to assess breath profile changes and correlation with endoscopy findings.
  Interventions: Diagnostic Test: Breath test
- Advanced Oesophageal cancer (T2/3/4): Patients who have been diagnosed with oesophageal adenocarcinoma attending hospital as part of their clinical care will be asked to give a breath sample prior to their endoscopy resection/ cancer operation.
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Patients will provide a breath test prior to gastroscopy or resection of Barrett's HGD lesion or oesophageal cancer.

SUMMARY:
This study aims to determine whether a breath test could be used for early detection of oesophageal cancer and Barrett's high grade dysplasia.

Patients who are attending for a planned gastroscopy or who are scheduled to undergo elective resection of histologically confirmed early stage oesophageal adenocarcinoma or dysplasia will be approached to provide a breath sample.

Multi platform mass spectrometry analysis will be performed to establish volatile biomarkers that can discriminate between early stage (T1) oesophageal cancer/ Hight grade dysplasia from non cancer healthy controls/non dysplastic Barrett's cancer.

DETAILED DESCRIPTION:
The incidence of oesophageal adenocarcinoma has been rising over the last decade. Despite improvements in oncological and surgical therapies the associated survival remains poor, mainly due to delays in diagnosis and advanced stage at presentation. Identifying patients at earlier stages as well as those at risk of cancer may lead to survival benefit. Barrett's oesophagus is an established risk factor for the development of oesophageal adenocarcinoma. It has an established histopathologic progression from low-grade, through high-grade dysplasia (HGD) to oesophageal adenocarcinoma (OAC). Barrett's oesophagus patients currently undergo regular endoscopic surveillance to allow earlier detection of oesophageal cancer.

The primary objective is to evaluate the diagnostic accuracy and clinical utility of the volatile organic compounds (VOC) in exhaled breath to detect early stage oesophageal adenocarcinoma and high-grade dysplastic Barrett's oesophagus.

All patients will be fasted for a minimum of 6 hours prior to the breath sample as part of their routine clinical care. Breath collection will be conducted using a previously validated method. Samples of breath (500ml) collected using "breath collecting device utilising bags". Breath samples collected within thermal desorption tubes (Markes International, Llantrisant, UK) will be transferred to a central laboratory for analysis by gas chromatography mass spectrometry (GC-MS) and proton transfer reaction time of flight mass spectrometry (PTR-ToF-MS). Raw data files will be extracted and analysed in accordance with established protocols.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and ≤90 years of age
* Undergoing gastroscopy or elective resection of histologically confirmed oesophageal adenocarcinoma/ high grade dysplasia
* Fasted >6 hours
* Able to provide informed written consent

Exclusion Criteria:

* Any patient <18 years or >90 years of age.
* Lacks capacity or is unable to provide informed written consent.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending for a planned gastroscopy as part of their Barrett's surveillance or under the two week wait rule or who are scheduled to undergo elective surgical or endoscopic resection of histologically confirmed early oesophageal adenocarcinoma/ high grade dysplasia will be eligible for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic accuracy of breath test for detection of early oesophageal cancer and Barrett's high grade dysplasia | 4 years
  Diagnostic accuracy will be measured by calculating the sensitivity and specificity of the test for detection of early oesophageal cancer/ high grade dysplasia. Sensitivity and specificity values are represented by a number between 0 to 1 indicating the test's ability to pick up true positive results and true negative results respectively, where a number closer to one indicates a greater detection ability.

SECONDARY OUTCOMES:
Diagnostic validation study of the breath profile for prediction of early oeosphageal cancer and high grade dysplasia | 3
  After diagnostic accuracy has been determined as per objective 1 by the discovery phase of the proposed study, a validation phase will then follow to confirm findings. Diagnostic accuracy of the validation phase results will be measured by calculating the sensitivity and specificity of the test for detection of T1 oesophageal cancer and dysplasia. Sensitivity and specificity values are represented by a number between 0 to 1 indicating the test's ability to pick up true positive results and true negative results respectively, where a number closer to one indicates a greater detection ability.

CONTACTS AND LOCATIONS:
Overall Officials: George B Hanna, FRCS PhD, Principal Investigator — Imperial College London
Locations (12):
- United Kingdom (12):
  - University Hospitals Birmingham Nhs Foundation Trust, Birmingham
  - University Hospital Dorset NHS Foundation Trust, Bournemouth
  - University Hospital Coventry and Warwickshire, Coventry
  - Royal Liverpool University Hospital, Liverpool
  - University College London Hospitals Nhs Foundation Trust, London
  - Guy'S and St Thomas' Nhs Foundation Trust, London
  - Imperial College Healthcare Trust, London
  - Newcastle Hospital NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Portsmouth Hospitals Nhs Trust, Portsmouth
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Betsi Cadwaladr University Health Board, Wrexham

IPD SHARING:
Plan to Share IPD: No